CLINICAL TRIAL: NCT04386564
Title: Prospective Parallel-Group Study of the Relationship Between Kidney Injury Severity and Severity of COVID-19
Brief Title: Kidney Injury Severity and COVID-19
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Other Study IDs: Sechenov-COVID19_AKI
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: COVID-19; Kidney Injury
Keywords: Coronavirus Infection; Kidney Function
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood,urine, sputum. Renal tissue only from post-portem kidney biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild COVID-19: Pneumonia without respiratory failure
  Interventions: Diagnostic Test: mRNA in urine test
- Moderate COVID-19 up to 60 years: Respiratory frequency ≥30/minute, blood oxygen saturation≤93%
  Interventions: Diagnostic Test: mRNA in urine test
- Moderate COVID-19 over 60 years old and severe COVID-19: Pneumonia with respiratory distress syndrome
  Interventions: Diagnostic Test: mRNA in urine test

INTERVENTIONS:
Diagnostic Test: mRNA in urine test — Assessment of renal function, expression of viral RNA in urine and assessment of radiological changes will be performed
  Other Names: chest and abdominal CT scan; CRP; Hb; Presepsin; eGFR; Ccr; UACR; UMA; Proteinuria

SUMMARY:
The authors hypothesize that the SARS-CoV-2 virus can affect the kidneys, causing them to be damaged. The present study aims to explain the mechanisms of kidney injury in patients diagnosed with COVID-19.

DETAILED DESCRIPTION:
In December 2019, an outbreak of the 2019 novel coronavirus disease (COVID-19) caused by the SARS coronavirus 2 (SARS-CoV-2) occurred in Wuhan, China. It has spread rapidly to other areas in China and worldwide. The most common manifestations of COVID-19 included fever, dry cough, dyspnea, myalgia, fatigue and radiographic evidence of pneumonia. Complications (acute respiratory distress syndrome, shock, acute cardiac injury, secondary infection, and acute kidney injury) and death may occur in severe cases. Recent reports showed that extrapulmonary symptoms (intestinal symptoms in 10-20% of patients) and renal failure in some patients may be associated with the interaction of the virus with angiotensin-converting enzyme 2 (ACE-2) receptors in other organs. It was suggested that ACE-2 expression in the kidneys can be the cause of kidney injury occurring in a number of patients with SARS-CoV-2.However, ACE-2 is not the only possible cause of kidney injury - sepsis-related cytokine storm can also lead to damage of kidney parenchyma.

The present study aims to explain the mechanisms of kidney injury in patients diagnosed with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia confirmed by CT scans

Exclusion Criteria:

* a history of chronic renal failure;
* a history of kidney transplantation;
* intake of substances with a history of renal toxicity (no later than a month before inclusion);
* patients with a single kidney;
* refusal of the patient to participate in the study;
* absence of SARS-CoV-2 virus smear from the nasopharynx in PCR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females with confirmed viral pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The effect of COVID-19 severity on the severity of renal failure | 2 months
  estimated glomerular filtration rate (eGFR), ml/min, in groups with mild, moderate and severe COVID-19

SECONDARY OUTCOMES:
The expression of viral RNA in the urine with the severity of renal failure | 2 months
  viral RNA concentration in urine, ME/ml
The severity of microalbuminuria in patients with COVID-19 of different conditions and renal failure | 2 months
  albumine excretion with urine, g/ml
Assessment of the severity of renal impairment in patients who died from COVID-19 | 2 months
  estimated glomerular filtration rate (eGFR), ml/min
Estimation of the duration of urinary viral RNA isolation in patients undergoing COVID-19 | 2 months
  Duration of viral RNA detection in urine by PCR, weeks
Expression of ACE-2 receptors in the kidneys of patients with renal failure who died from COVID-19 | 2 months
  expression of ACE-2 by imminohistochemistry at autopsy specimen

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, M.D., Ph.D., Principal Investigator — Sechenov University
Locations (1):
- Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No